CLINICAL TRIAL: NCT00671424
Title: An Evaluation of the Safety, Tolerability, and Pharmacodynamic Effects of GSK189075 When Administered With Furosemide or Hydrochlorothiazide
Brief Title: A Study To Compare Effects Of GSK189075 In Combination With Either Furosemide Or Hydrochlorothiazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KG2105251
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Interaction,; Diabetes,; healthy male subjects; GSK189075,; Diuretics,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Hydrochlorothiazide; remogliflozin etabonate; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydrochlorothiazide (HCTZ)
Drug: Remogliflozin etabonate (GSK189075)
Drug: Furosemide
  Other Names: Remogliflozin etabonate (GSK189075); Hydrochlorothiazide (HCTZ)

SUMMARY:
Many patients with type 2 diabetes also have conditions that are treated with diuretics. The patients may also be treated with GSK189075 for their diabetes. This study is planned to assess possible effects of administering GSK189075 in combination with two frequently used diuretics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male subjects who are between 18 and 50 years of age, inclusive.
* BMI within the range 19-30 kg/m2 (inclusive).
* Capable of providing signed and dated informed consent, which includes compliance with the requirements and restrictions listed in the consent form and with study-specific instructions provided by the site staff

Exclusion Criteria:

* Significant renal disease as manifested by one or more of the following:
* Symptoms of benign prostatic hyperplasia.
* Prostate-specific antigen level of greater than 10ng/mL (or equivalent to moderately elevated per the local lab).
* Any medical procedures requiring ingestion of radioactive agents within one week prior to dosing with study drug.
* Cholecystectomy within 6 months before the first scheduled dose of study drug.
* Any known or suspected gastrointestinal condition (or minor gastrointestinal surgery within 1 month prior to the first scheduled dose of study drug) that would likely interfere with the absorption or transit of study drug.
* Any subject with either documented cirrhosis or history consistent with a diagnosis of cirrhosis.
* History of gout.
* History of sensitivity to any of the study medications, or their components, which in the opinion of the investigator or GSK Medical Monitor, contraindicates participation.
* History of allergy to sulfonamides, sulfonylureas, carbonic anhydrase inhibitors, thiazides, loop diuretics (other than ethacrynic acid).
* Subjects with clinical laboratory values outside ranges specified in protocol at screening or Day 1:
* Significant ECG abnormalities at screening according to ranges specified in the protocol:
* Systolic/Diastolic blood pressure: less than 80/60 mmHg or greater than 150/95 mmHg at screening.
* Any clinically relevant abnormality identified on the screening physical or laboratory examination.
* Hemoglobin or hematocrit below the reference range at screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* The subject has a positive drug/alcohol test at screening or check in into the clinic. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months prior to screening.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study (whichever is longer): 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to latex

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Serum sodium and potassium concentrations: | baseline, Day 3, and Days 9-15

SECONDARY OUTCOMES:
adverse events: | each visit
Physical Exam: | screening,Days -1,15,follow-up
ECG & vital signs: | Days -1,3,8,9,14,15,follow-up
Clinical labs:screening: | Days -1,3,8-15,follow-up
blood pressure: | days 7,13
urine labs: | Days 7,8,9,13,14
weight: | Days -1,3,4,9,10,15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Columbus, Ohio, United States